CLINICAL TRIAL: NCT05165342
Title: Effectiveness and Safety of High Frequency Electrotherapy in Patients With Meibomian Gland Dysfunction : Randomized Controlled Trial
Brief Title: Effectiveness and Safety of High Frequency Electrotherapy in Patients With Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 845/63
Record Dates: First submitted 2021-11-17; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): This treatment is delivered by contact electrodes built in a mask, which is worn by the patient over closed eyes. The device setup is really easy and intuitive.
  Interventions: Device: Rexon-eye
- Sham-intervention (Sham Comparator): The same device as treatment but the power of device will be set to ZERO power.
  Interventions: Device: Rexon-eye

INTERVENTIONS:
Device: Rexon-eye — a technique in which low-intensity, high-frequency (a spectrum of frequencies ranging from 4 MHz to 64 MHz) electric currents are administered to a biological tissue through contact electrodes
  Other Names: Quantum Molecular Resonance device

SUMMARY:
This study is a prospective randomized double-masked sham-controlled clinical trial to determine the clinical improvement, safety and mechanism of action by evaluation inflammatory cytokine, and amount of bacteria and demodex, after high frequency electrotherapy or called quantum molecular resonance treatment in patients with meibomian gland dysfunction.

DETAILED DESCRIPTION:
The Rexon-eye is quantum molecular resonance device which was published in previous study that could treat meibomian gland dysfunction. Participants in this study will have Rexon-eye treatment at baseline (after recording of baseline characteristics and giving and inform consent), day 7, day 14, day 21. The evaluation for most parameter except for safety parameter will be recorded at baseline, 1 month after last treatment, and 2 mont after last treatment. Safety parameter will be recorded in all 4 follow-ups. During study, all participant will instructed to use same artificial tears for four time a day.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and sign an informed consent form
2. > 18years of age
3. Able and willing to comply with the treatment/follow-up schedule and requirements
4. Presence of meibomian gland on each lower eyelid's meibography
5. Current diagnosis of stage 1-4 of MGD in both eyes, according to the International Workshop on Meibomian Gland Dysfunction: Report of the Subcommittee on Management and Treatment of Meibomian Gland Dysfunction

Exclusion Criteria:

1. Contact lens wearer within the past 1 month and throughout the study
2. Recent ocular surgery or eyelid surgery within the past 6 months
3. Neuro-paralysis in the planned treatment area within the past 6 months
4. Current use of punctal plugs
5. Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
6. Uncontrolled infections or uncontrolled immunosuppressive diseases
7. Subjects who have undergone refractive surgery within the past 6 months
8. Patients who had ocular infection within 6 months
9. Pregnancy and lactation
10. Any condition revealed during the eligibility screening process whereby the physician deems the subject inappropriate for this study
11. Declared legally blind in one eye
12. Lipiflow treatment, or any equivalent treatments, within the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
non-invasive tear break-up time (NITBUT) | 1 month after last treatment (2 month from baseline)
  Change from baseline NITBUT at 1 month after last treatment
non-invasive tear break-up time (NITBUT) | 2 month after last treatment (3 month from baseline)
  Change from baseline NITBUT at 2 month after last treatment

SECONDARY OUTCOMES:
Ocular Surface Index Score scored (OSDI score) | 1 month after last treatment (2 month from baseline)
  Change from baseline OSDI score at 1 month after last treatment
Lid margin thickening grade | 1 month after last treatment (2 month from baseline)
  Change from baseline Lid margin thickening grade at 1 month after last treatment
Lid margin notching grade | 1 month after last treatment (2 month from baseline)
  Change from baseline Lid margin notching grade at 1 month after last treatment
Lid margin telangiectasia | 1 month after last treatment (2 month from baseline)
  Change from baseline Lid margin telangiectasia at 1 month after last treatment
meibomian gland cupping grade | 1 month after last treatment (2 month from baseline)
  Change from baseline meibomian gland cupping grade at 1 month after last treatment
Lid meibography grade (upper and lower lid) | 1 month after last treatment (2 month from baseline)
  Change from baseline Lid meibography grade at 1 month after last treatment
meibum expressibility grade | 1 month after last treatment (2 month from baseline)
  change from baseline meibum expressibility grade at 1 month after last treatment
meibum quality grade | 1 month after last treatment (2 month from baseline)
  Change from baseline meibum quality grade at 1 month after last treatment
Amount of bacteria culture from lid margin and meibum (colony forming unit) | 1 month after last treatment (2 month from baseline)
  Change from baseline meibum quality grade at 1 month after last treatment
Tear cytokine level (Interleukin-6, Interferon-gamma, Interleukin-1RA) | 1 month after last treatment (2 month from baseline)
  Change from baseline Tear cytokine level at 1 month after last treatment
Tear osmole | 1 month after last treatment (2 month from baseline)
  Change from baseline Tear osmole level at 1 month after last treatment
Schirmer test (not use anaesthesia, mm) | 1 month after last treatment (2 month from baseline)
  Change from baseline schirmer test at 1 month after last treatment
Tear meniscus height | 1 month after last treatment (2 month from baseline)
  Change from baseline Tear meniscus height at 1 month after last treatment
TFLLT (Tear film lipid layer thickness) | 1 month after last treatment (2 month from baseline)
  Change from baseline TFLLT at 1 month after last treatment
Bulbar conjunctiva hyperaemia (graded by Janvis score) | 1 month after last treatment (2 month from baseline)
  Change from baseline Bulbar conjunctiva hyperaemia at 1 month after last treatment
Corneal and conjunctiva staining score (Use fluorescent and lissamine green stain) | 1 month after last treatment (2 month from baseline)
  Change from baseline corneal and conjunctival stain at 1 month after last treatment
Incidence of adverse event | at every visit after treatment (baseline, day7, day14, day21)
  Incidence of adverse event
best spectacle corrected visual acuity (logMAR) | at every visit before treatment (baseline, day7, day14, day21)
  Any change from baseline best spectacle corrected visual acuity (logMAR) at day7, day14, and day 21
uncorrected visual acuity (logMAR) | at every visit before treatment (baseline, day7, day14, day21)
  Any change from baseline uncorrected visual acuity (logMAR) at day7, day14, and day 21
Ocular Surface Index Score scored (OSDI score) | 2 month after last treatment (3 month from baseline)
  Change from baseline OSDI score at 2 month after last treatment
Lid margin thickening grade | 2 month after last treatment (3 month from baseline)
  Change from baseline Lid margin thickening grade at 2 month after last treatment
Lid margin notching grade | 2 month after last treatment (3 month from baseline)
  Change from baseline Lid margin notching grade at 2 month after last treatment
Lid margin telangiectasia | 2 month after last treatment (3 month from baseline)
  Change from baseline Lid margin telangiectasia at 2 month after last treatment
meibomian gland cupping grade | 2 month after last treatment (3 month from baseline)
  Change from baseline meibomian gland cupping grade at 2 month after last treatment
Lid meibography grade (upper and lower lid) | 2 month after last treatment (3 month from baseline)
  Change from baseline Lid meibography grade at 2 month after last treatment
meibum expressibility grade | 2 month after last treatment (3 month from baseline)
  change from baseline meibum expressibility grade at 2 month after last treatment
meibum quality grade | 2 month after last treatment (3 month from baseline)
  Change from baseline meibum quality grade at 2 month after last treatment
Schirmer test (not use anaesthesia, mm) | 2 month after last treatment (3 month from baseline)
  Change from baseline schirmer test at 2 month after last treatment
Tear meniscus height | 2 month after last treatment (3 month from baseline)
  Change from baseline Tear meniscus height at 2 month after last treatment
TFLLT (Tear film lipid layer thickness) | 2 month after last treatment (3 month from baseline)
  Change from baseline TFLLT at 2 month after last treatment
Bulbar conjunctiva hyperaemia (graded by Janvis score) | 2 month after last treatment (3 month from baseline)
  Change from baseline Bulbar conjunctiva hyperaemia at 2 month after last treatment
Corneal and conjunctiva staining score (Use fluorescent and lissamine green stain) | 2 month after last treatment (3 month from baseline)
  Change from baseline corneal and conjunctival stain at 2 month after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lita Uthaithammarat, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
After submit to journal, I will send the raw data to the journal and published as supplementary file
Supporting Information: Study Protocol
Time Frame: After submitting to journal.
Access Criteria: I am happy to share all of my protocol and also my raw data to who which interested and plan to do the study about Recon-eye device. Moreover, If journal I have submitted want to publish all data and research protocol as supplementary or request me to upload in any data sharing website, I will follow their request.

REFERENCES:
- [Result] Ferrari G, Colucci A, Barbariga M, Ruggeri A, Rama P. High Frequency Electrotherapy for the Treatment of Meibomian Gland Dysfunction. Cornea. 2019 Nov;38(11):1424-1429. doi: 10.1097/ICO.0000000000002063. PMID 31356415